CLINICAL TRIAL: NCT02824328
Title: A Pilot Study Investigating the Effect of Chemotherapy on the Tumoral Immunoprofile of Gynecologic Cancers
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00066330; 5K12HD043446-14 (NIH)
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Uterine Endometrial Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood (30ml) on the day of biopsy
  2. Additional tissue at time of clinical biopsy (if it is safe for additional tissue to be collected during this time beyond what is clinically indicated, an effort will be made to do so. All biopsy tissue collected will be sent to pathology, including any additional tissue. Tissue remaining after pathology has performed their clinical care requirements will be collected) OR Collection of excess tissue at time of clinical biopsy (if it is unsafe for additional tissue to be collected, only tissue in excess of what is what pathology uses will be collected)
  3. Excess ascites at time of paracentesis (if performed for diagnostic/therapeutic purposes)
  4. Additional blood (30ml) within 3 days of surgery
  5. Excess tumor tissue and ascites at the time of cytoreductive surgery
  6. Blood (30ml) at the next scheduled visit after completion of post-surgical adjuvant therapy.
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to collect biologic samples (i.e. tumor tissue, ascites, and/or blood), from patients undergoing standard of care therapy for a gynecologic malignancy. To detect changes in the immune response following chemotherapy, collection of biologic samples will occur at baseline and at the time of surgery following chemotherapy.

DETAILED DESCRIPTION:
This is a single-institution, non-interventional prospective observational study allowing for specimen and data collection. All participants will receive standard of care surgery and chemotherapy, determined by the gynecologic oncologist and per institutional protocols. Patients with a presumed diagnosis of an eligible gynecologic malignancy (epithelial ovarian, fallopian tube, primary peritoneal, or uterine endometrial cancer) who are being considered for neoadjuvant chemotherapy prior to confirmatory biopsy will be given the option to enroll on this study.

Patients will undergo standard biopsy or endometrial curettage to confirm diagnosis. Additional tumor tissue for research purposes will be collected at the time of biopsy (if safely available). Patients who are undergoing diagnostic or therapeutic paracentesis will have the option to consent to allow excess ascites to be evaluated in this research protocol. Additionally, a research blood sample will be collected on the same day as the biopsy/curettage.

After confirmation of diagnosis, chemotherapy administration will proceed per standard institutional protocol and surgical planning will be performed by the treating gynecologic oncologist. Excess tumor tissue and ascites from the cytoreductive surgery will be collected for immune profiling. An additional vial of blood for research will be collected within 3 days prior to surgery. Post-surgical treatment and chemotherapy will proceed per standard procedures. After completion of post-surgical adjuvant therapy, an additional vial of blood for research will be collected (at next scheduled clinic visit).

ELIGIBILITY:
Inclusion Criteria:

1. Presumed diagnosis of tumor of müllerian origin, specifically epithelial ovarian, fallopian tube, primary peritoneal, or uterine endometrial cancer. After biopsy portion of study, only patients with histologically or cytologically confirmed diagnosis of eligible malignancies will continue.
2. Be considered a candidate for neoadjuvant chemotherapy per institutional standards.
3. Be willing and able to provide written informed consent for the trial.
4. Be ≥ 18 years of age on day of signing informed consent.
5. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen upon agreement of the investigator.
6. Have a performance status of 0-2 on the ECOG Performance Scale.
7. Female subjects of childbearing potential should have a negative urine pregnancy test within 48 hours prior initial biopsy or administration of chemotherapy whichever comes first.

Exclusion Criteria:

1. Is currently participating and receiving a study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device for this diagnosis.
2. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
3. Has a history or current evidence of any condition (i.e. infection), therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
4. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
5. Is pregnant or breastfeeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a presumed diagnosis of an eligible gynecologic malignancy (epithelial ovarian, fallopian tube, primary peritoneal, or uterine endometrial cancer) who are being considered for neoadjuvant chemotherapy prior to confirmatory biopsy will be given the option to enroll on this study.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2016-06; Primary Completion 2019-07-25 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Change in number and type of tumor infiltrating lymphocytes | baseline, post treatment (approximately 6 months)
  To assess changes in the immune response through the characterization of tumor infiltrating lymphocytes (TILs) after administration of chemotherapy. Biomarker testing is for the purpose of biological research and is not intended to test or develop an in-vitro diagnostic test.
Change in expression level of Inflammatory mediators | baseline, post treatment (approximately 6 months)
  To assess changes in immune response through the characterization of inflammatory mediators after administration of chemotherapy. Biomarker testing is for the purpose of biological research and is not intended to test or develop an in-vitro diagnostic test.
Change in tumor expression level of PD-L1 | baseline, post treatment (approximately 6 months)
  To assess changes in the immune response through the characterization of tumor expression of PD-L1 after administration of chemotherapy. Identify immune signatures/biomarkers that predict treatment outcomes. Biomarker testing is for the purpose of biological research and is not intended to test or develop an in-vitro diagnostic test.
Changes in HLA-type | baseline, post treatment (approximately 6 months)
  To assess changes in HLA-type after administration of chemotherapy. Identify immune signatures/biomarkers that predict treatment outcomes. Biomarker testing is for the purpose of biological research and is not intended to test or develop an in-vitro diagnostic test.

CONTACTS AND LOCATIONS:
Overall Officials: Angeles A Secord, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided